CLINICAL TRIAL: NCT06597578
Title: Prospektives KÖln Bonner Register Zur Extraktion Von Schrittmacher- Und ICD-Sonden (KÖBES)
Brief Title: Prospective Köln Bonn Registry for the Extraction of Pacmaker and ICD Leads
Acronym: KOBES
Status: Recruiting | Type: Observational
Sponsor: Evangelic Hospital Kalk Cologne (Other)
Responsible Party: Principal Investigator, Frank Eberhardt, Assistant Professor, Evangelic Hospital Kalk Cologne
Other Study IDs: 2023KÖB
Record Dates: First submitted 2024-02-21; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-02

CONDITIONS: Infections; Pacemaker, Artificial; Defibrillators, Implantable
Keywords: lead extraction; cardiac device; infection; complication; pacemaker; implantable cardioverter-defibrillator; extraction tools
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Extraction tools — The effect of different extraction tools on outcome parameters will be evaluated

SUMMARY:
The KOBES registry is an all-comers prospective clinical registry of the cooperative Köln Bonn lead extraction center. All patients undergoing complex lead extraction procedures (i.e. indwelling leads > 6months) in the hybrid operating room with cardiothoracic standby will be included in the registry. Preoperative, intraoperative/procedural and postoperative parameters will be recorded. All patients will be asked to provide written informed consent. Data will be pseudonomyzed and entered into a data sheet. Data will be monitored by a board and evaluated independently.

DETAILED DESCRIPTION:
The following parameters will be included in the registry Preoperative

General:

* pacemaker / ICD indication
* Ejektionsfraktion
* previous cardiac surgery / TAVR
* specific cardiac disease: IHD, CMP (DCM, HCM, andere), Primary electrical disease if ICD:
* primary / secondary prevention concomitant disease:HTN, DM
* CRF; GFR (ml/min)
* if yes: dialysis ?
* anticoagulation / antithrombotic therapy: Ja/Nein

Indication:

* infection (local/systemic), classification
* blood culture positive/negative
* swab positive
* classification
* TEE: pos/neg
* Device malfunction
* Phlebography y/n
* Vascular access y/n
* Number of Leads and Type
* uni/bipolar / age / abandoned leads
* ICD-leads: single-/dual-coil, age / abandoned leads

Intraoperative:

General:

* type of anaethesia
* TEE y/n
* Safety wire y/n
* temporary pacing wire y/n

Access:

* Subclavia r/l/bil
* Femoral: y/n; if yes: planned / Bailout: geplant Tools
* LLD: y/n; Number
* Mechanical sheath and type
* Laser sheath
* Additional tools: Loop-Snare / Needle-Eye Snare / Rat-Tooth Result : extraction: complete / partial / failed
* procedural success: y/n
* infection: procedural / clinial success
* Safety lead y/n
* temporary pacing wire in situ Intraoperative complications
* vascular injury
* pericardial effusion / tamponade
* pericardiocentesis
* occlusion ballon
* thoracotomy
* Intraoperative catecholamines
* death

Postoperative:

* duration
* hospital stay
* postoperative active system
* transvenous / epicardial / capsule/ subcutaneous / extravascular
* type of pacemaker
* type of ICD
* Wenn ja: transvenös / subkutan

Postoperative complications:

* hematoma / seroma / fistula
* further interventions: Revision / hematoma/ reinfection

ELIGIBILITY:
Inclusion Criteria:

* All patients with a standard indication for lead extraction according to the HRS / EHRA guidelines

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting at the Koeln Bonn cooperative lead extraction center for a complex lead extraction
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedural success | 1 week
  Complete / partial success with combined femoral superior extraction compared to superior extraction only

SECONDARY OUTCOMES:
Complications | 1 year
  Periprocedural complications

CONTACTS AND LOCATIONS:
Overall Officials: Frank Eberhardt, MD, Principal Investigator — EVKK
Locations (1):
- EVKK, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No